CLINICAL TRIAL: NCT04508712
Title: Long-term Outcomes in Patients With COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: COVID-19 Prognosis
Record Dates: First submitted 2020-08-08; First posted 2020-08-11 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: COVID-19
Keywords: COVID-19; long-term outcomes
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Long-term outcomes from coronavirus disease 2019 (COVID-19) are currently unknown. This study will collect daily living status of survivors of COVID-19.

DETAILED DESCRIPTION:
The ongoing pandemic of coronavirus disease 2019 (COVID-19), due to the newly discovered severe acute respiratory syndrome coronavirus 2 (SAR-CoV-2), has caused a worldwide increase in hospitalization for pneumonia with multi- organ disease. Survival from sepsis is associated with increased risk for mortality for at least 2 years. Therefore, substantial sequelae including new physical disability, new cognitive impairment and increased vulnerability to further health deterioration are likely to be seen in survivors of COVID-19. The investigators conduct this study to investigate daily living status of survivors of COVID-19 using telephone interview questionnaire including Activity Daily Living(ADL), modified Medical Research Council(mMRC),modified Telephone Interview for Cognitive Status (TICS-m), Zung Self-rating Depression Scale(SDS), Carcinologic Handicap Index (CHI), and New York Heart Association (NYHA) functional class.

ELIGIBILITY:
Inclusion Criteria:

* Survivors who had been admitted in Leishenshan Hospital for COVID-19 patients in Wuhan, China

Exclusion Criteria:

* Patients who were < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll survivors of COVID-19 aged over 18 years old who had been admitted in Leishenshan Hospital for COVID-19 patients in Wuhan, China.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Physical functions | 4-6 months
  Physical functions will be assessed using Activities of daily living (ADL) scale. Minimum value:0, Maximum value: 100. Higher scores mean a better outcome.
Respiratory function | 4-6 months
  Respiratory function will be assessed using modified Medical Research Council(mMRC) scale. Minimum value:0, Maximum value: 4. Higher scores mean a worse outcome.
Cognitive function | 4-6 months
  Cognitive function will be assessed using modified Telephone Interview for Cognitive Status (TICS-m) scale. Minimum value:0, Maximum value: 50. Higher scores mean a better outcome.
Depression status | 4-6 months
  Depression status will be assessed using Zung Self-rating Depression Scale(SDS). Minimum value:25, Maximum value: 125. Higher scores mean a worse outcome.
Sensory functions | 4-6 months
  Sensory functions will be assessed using Carcinologic Handicap Index (CHI). Minimum value:0, Maximum value: 144. Higher scores mean a worse outcome.
Heart function | 4-6 months
  Heart function will be assessed using New York Heart Association (NYHA) functional class. Minimum value:1, Maximum value: 4. Higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Yu, MD,PhD, Study Director — Renji Hospital, School of Medicine, Shanghai Jiaotong University, China
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Pudong, Shanghai Municipality, China